CLINICAL TRIAL: NCT01288664
Title: Efficacy and Safety of Tacrolimus Sustained-release Capsules in Induction Phase Treatment in Lupus Nephritis
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: sponsor withdraw from this study
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Xueqing Yu, Sun Yat-sen University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSU-PRGLN-002
Record Dates: First submitted 2011-02-01; First posted 2011-02-02 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2013-12

CONDITIONS: Lupus Nephritis
Keywords: Lupus Nephritis; Tacrolimus; Induction Phase
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ADVAGRAF (Experimental): Tacrolimus Sustained-release Capsules (ADVAGRAF) treatment in induction phase for 6 months
  Interventions: Drug: ADVAGRAF

INTERVENTIONS:
Drug: ADVAGRAF — Tacrolimus Sustained-release Capsules (ADVAGRAF) Started: 0.05-0.1mg/kg/d, one time per day, the blood level:5-10ng/ml in induction phase.
  Other Names: ADVAGRAF:Tacrolimus Sustained-release Capsules

SUMMARY:
This is a pilot study to evaluate the efficacy and safety of Tacrolimus Sustained-release Capsules (ADVAGRAF) for the induction therapy of Lupus Nephritis (LN) (V, III +V, IV+V).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of either sex, 14-65 years of age;
2. Diagnosis of systemic lupus erythematosus (SLE) according to the albumin-creatinine ratio (ACR) criteria (1997);
3. Kidney biopsy within the 6 months prior to study with a histologic diagnosis (ISN/RPS 2003 classification of LN) class V, III +V, IV+V;
4. LN (Class IV+V): proteinuria > 1g/24hr or Scr > 1.3 mg/dl or active urinary sediment (erythrocyte cast, > 5 white blood cell count (WBC) /high power field (hpf)(excluding infection ), > 5 red blood cell count (RBC)/hpf;
5. LN (Class V or III +V ): proteinuria > 2g/24hr or Scr > 1.3 mg/dl;
6. Provision of written informed consent by subject or guardian

Exclusion Criteria:

1. Inability or unwillingness to provide written informed consent
2. Usage of immunosuppression therapy (MMF, Cyclophosphamide (CTX), Cyclosporine A (CysA), methotrexate (MTX) ect) for more than 1 week within 1 month or Pulse intravenous MP treatment prior to recruitment
3. Scr > 4mg/dl (354umol/L)
4. Needing pulse intravenous Methylprednisolone (MP) or intravenous immunoglobulin
5. Lupus encephalopathy
6. Diagnosed diabetes mellitus (DM); Malignant tumors (except fully cured basal cell carcinoma)
7. History of significant gastrointestinal disorders (e.g. severe chronic diarrhea or active peptic ulcer disease) within 3 month prior to enter this study
8. Any Active systemic infection or history of serious infection within one month of entry
9. known infection with HIV, hepatitis B, or hepatitis C
10. Known hypersensitivity or contraindication to tacrolimus, corticosteroids
11. Participation in another clinic trial and/or receipt of investigational drugs within 4 weeks prior to screening
12. Pregnancy, nursing or use of a non-reliable method of contraception.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Remission rate (complete or partial remission) | 6 months

SECONDARY OUTCOMES:
proteinuria | every 3 months,up to 6 months
Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) scores | every 3 months, up to 6 months
  SLEDAI (Systemic Lupus Erythematosus Disease Activity Index, Bombardier et al, 1992).
Number of participants with adverse events as a measure of safety and tolerability | every 3 months, up to 6 months
  Adverse events,including infections, transient increases in serum creatinine, gastrointestinal complaints, liver function disorder and glucose intolerance, etc.
renal function | every 3 months, up to 6 months
relapse | every 3 months, up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yu Xueqing, MD, Principal Investigator — Department of Nephrology, 1st Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China